CLINICAL TRIAL: NCT02513693
Title: Effect of Deep Neuromuscular Blockade on Surgical Conditions and Recovery After Robotic Radical Prostatectomy: a Prospective Randomized Study
Brief Title: Deep Neuromuscular Blockade During Robotic Radical Prostatectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Palacky University (Other)
Collaborators: University Hospital Olomouc (Other); Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Milan Adamus, MD, PhD, MBA, Milan Adamus, MD, PhD, MBA, Palacky University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGA_LF_2015_012
Record Dates: First submitted 2015-07-28; First posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Neuromuscular Blockade
Keywords: Anesthesia; Rocuronium; Sugammadex; Neostigmine; TOF; Radical Prostatectomy; Robotic Surgery; Accelerometry
MeSH Terms: interventions — Rocuronium; Neostigmine; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Neuromuscular Blockade (Experimental): Drug: rocuronium + neostigmine
  Administration of rocuronium 0,6 mg/kg iv, top-ups 5-10 mg iv to target value of Train-of-Four (TOF) count = 1-2, TOF-count measurement every 1 min. Neuromuscular blockade reversal at the end of anesthesia: neostigmine 0.03 mg/kg iv + atropine 0.5-1.0 mg iv Induction of anesthesia: midazolam 1-2 mg iv, sufentanil 10-30 mcg iv, propofol 1.5-2.5 mg/kg iv Anesthesia: sevoflurane in air to target 1.2-1.5 minimal alveolar concentration (MAC). Rescue medication: sevoflurane, propofol 20-40 mg iv Extubation when patient is conscious and attained the recovery from neuromuscular blockade to a TOF-ratio of at least 0,9.
  Interventions: Drug: Standard neuromuscular blockade
- Deep Neuromuscular Blockade (Experimental): Drug: rocuronium + sugammadex
  Administration of rocuronium 0,6 mg/kg iv, top-ups 5-10 mg iv to target value of Post-tetanic Count (PTC) = 1-2; PTC measurement every 4 min. Neuromuscular blockade reversal at the end of anesthesia: sugammadex 2 mg/kg iv (when PTC is 18-20 and TOF-count 0) or sugammadex 4 mg/kg iv (when PTC under 18).
  Induction of anesthesia: midazolam 1-2 mg iv, sufentanil 10-30 mcg iv, propofol 1,5-2,5 mg/kg iv Anesthesia: sevoflurane in air to target 1.2-1.5 minimal alveolar concentration (MAC). Rescue medication: sevoflurane, propofol 20-40 mg iv.
  Extubation when patient is conscious and attained recovery from neuromuscular blockade to a TOF-ratio of at least 0,9.
  Interventions: Drug: Deep neuromuscular blockade

INTERVENTIONS:
Drug: Standard neuromuscular blockade — Standard neuromuscular block provided by rocuronium to TOF-count 1-2. Reversal of the block with neostigmine.
  Other Names: Rocuronium + neostigmine
  Arms: Standard Neuromuscular Blockade
Drug: Deep neuromuscular blockade — Deep neuromuscular block provided by rocuronium to PTC 1-2. Reversal of the block with sugammadex.
  Other Names: Rocuronium + sugammadex
  Arms: Deep Neuromuscular Blockade

SUMMARY:
Basic requirement for safe performance of the robotic intra-abdominal surgery is a calm and clear surgical field after the introduction of a capnoperitoneum. That can be enabled by a neuromuscular blockade. Provision of standard neuromuscular blockade is a compromise between optimal surgical conditions (sufficiently deep block) and capability to antagonize the block rapidly at the end of the surgery. With rocuronium, it is possible to maintain deep neuromuscular blockade safely until the very end of the surgery, and unlike with spontaneous recovery or reversal of the block with neostigmine, administration of sugammadex at the end of the surgery will enable quick and consistent reversal of the block. Project is focused on comparison of the parameters of deep and standard neuromuscular blockade - surgical conditions (primary endpoint), quality of recovery and turnover time (secondary endpoints).

DETAILED DESCRIPTION:
Balanced anesthesia is an anesthetic procedure of choice for intra-abdominal surgery. Main components of this procedure are loss of consciousness, treatment of pain and appropriate neuromuscular blockade (NMB). Peripheral neuromuscular blocking agents (NMBA) are drugs used for muscle relaxation during balanced anesthesia. Their use plays essential role for tracheal intubation, orotracheal tube tolerance, introduction of mechanical ventilation and provision of calm surgical field.

In laparoscopic procedures, introduction of capnoperitoneum for good visibility in surgical field is necessary. From anesthetic point of view this requirement can be met by adequate muscle relaxation. After withdrawal of capnoperitoneum at the end of the surgery the procedure is usually terminated quickly (this phase consists only from suture of a peritoneum and the small incisions through which instruments were inserted). Spontaneous recovery from NMB or usual reversal of the block by neostigmine are not fast and reliable enough at this moment. During standard neuromuscular blockade the dosage of NMBA is a compromise between optimal surgical conditions (sufficiently deep block) and capability to antagonize the block rapidly at the end of the surgery. Introduction of sugammadex into clinical praxis brings the potential to change this paradigm. With rocuronium, it is possible to maintain deep neuromuscular blockade safely until the very end of the surgery and unlike with spontaneous recovery or reversal of the block with neostigmine, administration of sugammadex at the end of the surgery will enable quick and consistent reversal of the block. Data about routine use of the deep block are rare, PubMed lists with search strategy [(deep neuromuscular blockade) AND (laparoscopic surgery OR laparoscopy)] 11 references (January 12, 2015, www.pubmed.com).

Patients undergoing robotic radical prostatectomy will be randomized to two groups differing in muscle relaxation strategy (standard vs. deep) and the type of antagonizing drug at the end of the surgery (neostigmine vs. sugammadex). Relevant end-points and the differences between groups with deep and standard neuromuscular blockade will be compared. Indication and dosage of rocuronium, neostigmine and sugammadex correspond to manufacturers' recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Informed consent
* Elective robotic radical prostatectomy
* American Society of Anesthesiologists (ASA) status 1-3

Exclusion Criteria:

* Age under 18 years
* American Society of Anesthesiologists (ASA) status over 3
* Indication for rapid sequence induction, signs of difficult airway severe neuromuscular, liver or renal disease
* Known allergy to drugs used in the study
* Malignant hyperthermia (medical history)

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Surgical condition | Every 15 minutes during surgery until final suture
  Surgical rating score (SRS) - surgical condition will be evaluated by surgeon every 15 minutes on predefined five point scale (excellent - above average - average - below average - poor). For each patient, the final score will be the average of all 15 min SRS values.

SECONDARY OUTCOMES:
Quality of recovery | 2 months
  Speed of clinical recovery by using Post-Operative Quality Recovery Scale (www.pqrsonline.org). PQRS will be evaluated at following time points:
  preoperatively, day (D) 1, D3, D7, month (M) 1, M2.
"Ready to leave operating room (OR)" time | Period of patient's presence at OR
  "Ready to leave OR time" will be defined as a time period (in minutes) from the time point of completing surgery to the time point, when patient is ready to leave OR to the facility providing postanesthesia care.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Adamus, MD,PhD,MBA, Study Director — Department of Anesthesiology and Intensive Care Medicine Palacky University Olomouc Faculty of Medicine and Dentistry; Vladimir Cerny, MD,PhD,FCCM, Principal Investigator — J. E. Purkinje University, Masaryk Hospital, Usti nad Labem, Czech Republic, Dept. of Anesthesiology, Perioperative Medicine and Intensive Care
Locations (2):
- Czechia (2):
  - Dept. of Anesthesiology and Intensive Care Medicine, University Hospital Olomouc, Olomouc
  - Dept. of Anesthesiology, Perioperative Medicine and Intensive Care, J. E. Purkinje University, Masaryk Hospital, Ústí nad Labem

REFERENCES:
- [Result] Lindekaer AL, Halvor Springborg H, Istre O. Deep neuromuscular blockade leads to a larger intraabdominal volume during laparoscopy. J Vis Exp. 2013 Jun 25;(76):50045. doi: 10.3791/50045. PMID 23851450
- [Result] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Gatke MR. Optimized surgical space during low-pressure laparoscopy with deep neuromuscular blockade. Dan Med J. 2013 Feb;60(2):A4579. PMID 23461992
- [Result] Boon M, Martini CH, Aarts LP, Bevers RF, Dahan A. Effect of variations in depth of neuromuscular blockade on rating of surgical conditions by surgeon and anesthesiologist in patients undergoing laparoscopic renal or prostatic surgery (BLISS trial): study protocol for a randomized controlled trial. Trials. 2013 Mar 1;14:63. doi: 10.1186/1745-6215-14-63. PMID 23452344
- [Result] Ding L, Zhang H, Mi W, Sun L, Zhang X, Ma X, Li H. [Effects of carbon dioxide pneumoperitoneum and steep Trendelenburg positioning on cerebral blood backflow during robotic radical prostatectomy]. Nan Fang Yi Ke Da Xue Xue Bao. 2015 May;35(5):712-5. Chinese. PMID 26018268
- [Result] Ding L, Zhang H, Mi W, He Y, Zhang X, Ma X, Li H. [Effects of dexmedetomidine on recovery period of anesthesia and postoperative cognitive function after robot-assisted laparoscopicradical prostatectomy in the elderly people]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2015 Feb;40(2):129-35. doi: 10.11817/j.issn.1672-7347.2015.02.003. Chinese. PMID 25769330
- [Result] Dogra PN, Saini AK, Singh P, Bora G, Nayak B. Extraperitoneal robot-assisted laparoscopic radical prostatectomy: Initial experience. Urol Ann. 2014 Apr;6(2):130-4. doi: 10.4103/0974-7796.130555. PMID 24833824
- [Result] Kopman AF, Naguib M. Laparoscopic surgery and muscle relaxants: is deep block helpful? Anesth Analg. 2015 Jan;120(1):51-58. doi: 10.1213/ANE.0000000000000471. PMID 25625254
- [Result] Donati F, Brull SJ. More muscle relaxation does not necessarily mean better surgeons or "the problem of muscle relaxation in surgery". Anesth Analg. 2014 Nov;119(5):1019-21. doi: 10.1213/ANE.0000000000000429. No abstract available. PMID 25329018
- [Result] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Result] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Lindekaer AL, Riber C, Gatke MR. Surgical space conditions during low-pressure laparoscopic cholecystectomy with deep versus moderate neuromuscular blockade: a randomized clinical study. Anesth Analg. 2014 Nov;119(5):1084-92. doi: 10.1213/ANE.0000000000000316. PMID 24977638
- [Result] Dubois PE, Putz L, Jamart J, Marotta ML, Gourdin M, Donnez O. Deep neuromuscular block improves surgical conditions during laparoscopic hysterectomy: a randomised controlled trial. Eur J Anaesthesiol. 2014 Aug;31(8):430-6. doi: 10.1097/EJA.0000000000000094. PMID 24809482
- [Result] Vijayaraghavan N, Sistla SC, Kundra P, Ananthanarayan PH, Karthikeyan VS, Ali SM, Sasi SP, Vikram K. Comparison of standard-pressure and low-pressure pneumoperitoneum in laparoscopic cholecystectomy: a double blinded randomized controlled study. Surg Laparosc Endosc Percutan Tech. 2014 Apr;24(2):127-33. doi: 10.1097/SLE.0b013e3182937980. PMID 24686347
- [Result] Gurusamy KS, Vaughan J, Davidson BR. Low pressure versus standard pressure pneumoperitoneum in laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 18;2014(3):CD006930. doi: 10.1002/14651858.CD006930.pub3. PMID 24639018
- [Result] Royse CF, Newman S, Chung F, Stygall J, McKay RE, Boldt J, Servin FS, Hurtado I, Hannallah R, Yu B, Wilkinson DJ. Development and feasibility of a scale to assess postoperative recovery: the post-operative quality recovery scale. Anesthesiology. 2010 Oct;113(4):892-905. doi: 10.1097/ALN.0b013e3181d960a9. PMID 20601860